CLINICAL TRIAL: NCT00001859
Title: Screening Protocol for Patients Needing a Kidney, Kidney-Pancreas, or Islet Cell Transplant
Brief Title: Screening for Patients Needing Kidney, Kidney-Pancreas, or Islet-Cell Transplant
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990120; 99-DK-0120
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-05-30

CONDITIONS: Diabetes Mellitus; Kidney Failure
Keywords: Evaluation; Diabetes; Renal Failure
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency

SUMMARY:
Kidney transplantation is the preferred treatment for most end-stage kidney disease. This procedure is limited, however, by two major factors: 1) a shortage of donor organs and 2) organ rejection by the recipient. The National Institute of Diabetes and Digestive and Kidney Diseases is screening patients with kidney failure or diabetes who may be eligible for kidney, kidney and pancreas, or islet cell transplantation.

Patients in this screening study are not offered treatment. When the screening is complete, patients will be offered an opportunity to participate in another institute study, or, if there are no active studies appropriate for the patient, other options will be suggested to the primary or referring physician. Patients found eligible for a study are not obligated to participate.

Screening for all patients typically consists of blood tests, urinalysis, electrocardiogram, PPD tuberculosis screen and pregnancy test. Chest and kidney X-rays and other studies may be done on patients determined eligible for a particular study, including transplantation. A summary of all test results will be sent to the referring physician unless the patient requests otherwise.

...

DETAILED DESCRIPTION:
This protocol is designed for screening of patients with renal failure and/or diabetes who may be eligible for kidney, kidney-pancreas, or islet cell transplantation. Its purpose is to allow detailed investigation into the renal and endocrine function of these patients, and the status of other organ systems that would determine their ability to safely tolerate specific aspects of other therapeutic research protocols. After completion of this screening process, the patient will either be offered a chance to participate in an active treatment protocol, or if no appropriate protocol is identified, will have recommendations for other treatment options relayed to the primary or referring physicians.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be entered on this protocol at the time of their first visit to the NIH Clinical Center Outpatient Clinic or Inpatient Services if:

The patient carries the diagnosis of a disorder for which the Transplant Branch has active research interest, and based on information received from an outside physician, they meet preliminary eligibility criteria for other specific research protocols.

The patient or the patient's guardian is capable of providing informed consent, and signs the informed consent after initial counseling by clinical staff. Separate consent forms for all interventional procedures will be obtained after explanation of the specific procedure.

EXCLUSION CRITERIA:

History of known malignancies except basal cell carcinoma of the skin.

Inability to give legal informed consent by self or legal guardian.

Inability or willingness to comply with protocol monitoring and therapy, including, among others, a history of noncompliance, circumstances where compliance with protocol requirements is not feasible due to living conditions, travel restrictions, access to urgent medical services, or access to anti-rejection drugs after the research protocol is completed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 1999-06-04; Study Completion 2014-05-30

CONTACTS AND LOCATIONS:
Overall Officials: Monique E Cho, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Peacock M, Bilezikian JP, Bolognese MA, Borofsky M, Scumpia S, Sterling LR, Cheng S, Shoback D. Cinacalcet HCl reduces hypercalcemia in primary hyperparathyroidism across a wide spectrum of disease severity. J Clin Endocrinol Metab. 2011 Jan;96(1):E9-18. doi: 10.1210/jc.2010-1221. Epub 2010 Oct 13. PMID 20943783